CLINICAL TRIAL: NCT05220059
Title: Effect of Polyphenol Extract on Cardiovascular Health Markers: a 4 Way Randomised Crossover Study
Acronym: Activ Acute
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Collaborators: University of Parma (Other); Activ'inside (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: REC/21/0029
Record Dates: First submitted 2021-11-26; First posted 2022-02-02 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Diseases; Endothelial Dysfunction; Blood Pressure
Keywords: Polyphenols; Cardiovascular Disease; Endothelial Function; Flow Mediated Dilation
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Polyphenols

STUDY DESIGN:
Intervention Model Description: Double-blind placebo controlled dose-response crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Polyphenol extract low dose (Experimental): 156mg single dose
  Interventions: Dietary Supplement: Polyphenol extract
- Polyphenol extract medium dose (Experimental): 222mg single dose
  Interventions: Dietary Supplement: Polyphenol extract
- Polyphenol extract high dose (Experimental): 333mg single dose
  Interventions: Dietary Supplement: Polyphenol extract
- Placebo (Placebo Comparator): Maltodextrin single dose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Polyphenol extract — Single dose
  Arms: Polyphenol extract high dose; Polyphenol extract low dose; Polyphenol extract medium dose
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
Endothelial dysfunction is an early predictor of cardiovascular events in at-risk patients. It is characterized by impaired endothelium-dependent dilation and is primarily caused by reduced nitric oxide bioavailability secondary to oxidative stress and inflammation. Finding dietary/dietary supplement-oriented approaches to improving endothelial function is of public health interest.

A randomized double-blind placebo controlled 4-way crossover study will be conducted to determine if acute consumption of a proprietary polyphenol extract (156 mg / 222 mg / 333 mg) will have a dose dependent response on endothelium-dependent flow-mediated dilation (ED-FMD) in fasting conditions, in comparison to a placebo (maltodextrin) in male smokers (20 - 45 years; n=20).FMD and blood pressure will be assessed at 0 & 2 hour timepoints following consumption of a single dose of polyphenol extract, accompanying blood samples will be collected to assess a range of endpoints including nitric oxide metabolites, angiotensin and polyphenols metabolites. Endothelium-independent vasodilation will also be measured 2 hours post consumption.

ELIGIBILITY:
Inclusion Criteria:

* At least two of the following risk markers; a BMI 25-30, waist circumference >94 cm, high normal blood pressure defined as either systolic 85-89 mmHg or diastolic 130-139 mmHg and have a normal ECG.

Exclusion Criteria:

* An individual who has tested positive (self reported) 2 weeks before the study period.
* A COVID-19 vaccinated individual who while receive the 1st or 2nd dose or booster 2 weeks before V0 or during the study period, due to the potential interaction of vaccine on markers assessed

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Polyphenols have a gender effect, a single sex population was chosen to increase homogeneity of test population and therefore likelihood of observing an FMD response. Males were selected.
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Flow Mediated Dilation | Change over 2 hours post dose
  Acute change in endothelium-dependent flow-mediated dilation

SECONDARY OUTCOMES:
Endothelium-independent vasodilation | Change after 2 hours post dose
  Acute change in endothelium-independent vasodilation in response to Glyceryl trinitrate (GTN) drug
Systolic blood pressure | Change over 2 hours post dose
  Measured by brachial cuff
Diastolic blood pressure | Change over 2 hours post dose
  Measured by brachial cuff

OTHER OUTCOMES:
Lipid profile | Visit 1, 0 hour only
  Measured in serum
Glucose | Visit 1, 0 hour only
  Measured in plasma
Tolerance and acceptability of extract | Immediately after each intervention
  Safety parameter. Measured on a 3-point likert scale (a lower value being a better outcome: 1, totally acceptable - 3, not at all acceptable)
Height | Visit 1, 0 hour only
  Measured in metres
Weight | 0 hour, at each time-point
  Measured in kg
Angiotensin-converting enzyme (ACE) | Change over 2 hours
  Exploratory outcome
Circulating polyphenol metabolites | Change over 2 hours
  Exploratory outcome. Measured in plasma
Endothelin1 | Change over 2 hours
  Exploratory outcome. Measured in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No